CLINICAL TRIAL: NCT04255394
Title: A Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data on the Exceed ABT Acetabular Cementless Cup System (Implants and Instruments)
Brief Title: Exceed ABT Acetabular Cup Cementless System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETEU.CR.EU37
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Correction of Functional Deformity
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Post-market Clinical Follow-up Study to provide safety, performance and clinical benefits data on the Exceed ABT acetabular cup (implants and instruments) when used in combination with ceramic liners or polyethylene articulating liners bearing Options.

A single-center, cohort observational clinical outcomes study

DETAILED DESCRIPTION:
Study Aim: To collect survivorship and clinical outcomes long-term data confirm-ing safety, performance and clinical benefits of the Exceed ABT ce-mentless cup when used in combination with ceramic and polyeth-ylene articulating liners

Objectives: Primary Objectives:

Clinical performance - as measured by clinical score data (HHS, WOMAC and Oxford Hip Score), radiographic as-sessments and survivorship which will be based on removal of the device.

Secondary Objectives:

Safety will be evaluated by monitoring incidence of adverse events. Length of study: 13 years (3 years enrollment plus 10 years follow-up): Post-operative follow-up visits at: 1, 3, 5, 7 and 10 years

ELIGIBILITY:
Inclusion Criteria:

* Patients who are capable of understanding the doctor's explanations, following his instructions and are able to participate in the follow-up program
* Patient who gave verbal consent to take part in the study at study commencement and written consent retrospectively at 10 years follow-up by signing the informed consent form according to the General data protection Regulation (GDPR) Patient Consent Form"
* Age: => 18 years
* Male and Female
* Non- inflammatory degenerative joint disease including osteoarthritis, avascular necrosis & post traumatic arthritis
* Rheumatoid arthritis,
* Correction of functional deformity
* Revision of failed joint reconstruction or treatment
* Treatment of femoral neck and trochanteric fractures of the proximal femur with femoral head involvement and which are unmanageable using other techniques

Exclusion Criteria:

* Infection, sepsis, and osteomyelitis
* Patients who are unwilling or unable to give consent, or to comply with the follow-up program
* The patient is known to be pregnant or breastfeeding
* Any vulnerable subjects (= individuals whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate)
* Uncooperative patient or patient with neurologic disorders who are incapable of fol-lowing instruction
* Osteoporosis
* Metabolic disorder which may impair bone formation
* Osteomalacia
* Local and distant foci of infection
* Rapid joint destruction, marked bone loss or bone resorption apparent on roent-genogram
* Vascular insufficiency, muscular atrophy, or neuromuscular disease
* Skeletal immaturity
* Morbid obesity
* Foreign body sensitivity. Where suspected, material sensitivity tests are to be made prior to implantation
* Any condition that may interfere with the survival of the implant such as Paget's disease, Charcot's disease, sickle cell anaemia or traits, lower extremity muscular atrophy or neuromuscular disease'

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Female ≥18 years
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-31 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A MoP: Exceed ABT cup with Cobalt Chrome head Ringloc-X poly Liner (called MOP, metal on Poly)
- Group B CoC: Exceed ABT cup with Ceramic head and ceramic Liner (called CoC, ceramic on ceramic)
Period: Overall Study
Arm/Group | Group A MoP | Group B CoC
Started | 220 | 457
Treated | 208 | 449
Completed | 38 | 138
Not Completed | 182 | 319
Not completed — Death | 35 | 25
Not completed — Device removed | 2 | 10
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Screen Failure/Not treated | 12 | 8
Not completed — Lost to Follow-up | 123 | 265
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A MoP | Group B CoC | Total
Number analyzed (Participants) | 220 | 457 | 677
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (5.6) | 61.0 (9.3) | 65.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 284 | 409
  Male | 95 | 173 | 268
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 220 | 457 | 677
Operative Side [Count of Participants; unit: Participants]
  Right | 127 | 238 | 365
  Left | 93 | 219 | 312
Diagnosis [Count of Participants; unit: Participants]
  Osteoarthritis | 209 | 411 | 620
  Other | 11 | 46 | 57

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Score
Description: Clinical performance - as measured by clinical score data (HHS). The HHS was developed for the assessment of the results of hip surgery, and is intended to evaluate various hip disabilities and methods of treatment in an adult population. The domains covered are pain, function, absence of deformity, and range of motion. The score has a minimum of 0 and a maximum of 100 points.
  The scale: Excellent:90 - 100, Good: 80 - 89, Fair: 70 - 79, Poor: < 70.
Time Frame: 10 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A MoP | Group B CoC
Number analyzed (Participants) | 28 | 134
score on a scale | 89.8 (11.2) | 90.4 (13.2)

2. Primary Outcome: Western Ontario and McMasters Universities Osteoarthritis Index-WOMAC Pain Score
Description: Clinical performance - as measured by clinical score data - womac pain The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties The scores for each subscale are summed up, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for physical function. A higher score indicates a worse clinical outcome.
  Womac pain score is reported here.
Time Frame: 10 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A MoP | Group B CoC
Number analyzed (Participants) | 38 | 148
score on a scale | 6.1 (2.5) | 6.8 (3.5)

3. Primary Outcome: 10 Year Survivorship
Description: Calculated Kaplan-Meier Survivorship based on revision of any component for any reason. Presented as the % of participants with the implant still in place 10 years post-operative.
Time Frame: 10 years post-operative
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group A MoP | Group B CoC
Number analyzed (Participants) | 208 | 449
percentage of participants | 90.47 [84.61 to 96.33] | 97.32 [95.42 to 99.23]

4. Secondary Outcome: Oxford Hip Score
Description: The Oxford hip score (OHS) is self-completion patient-centered outcome measure tool designed to assess disability in patients undergoing total hip replacement. The OHS consists of 12 questions about pain and disability experienced over the past four weeks. Each item has five response categories, given a score of between 1-5 (low disability to high disability). Scoring involves summating the total for each item to produce a final score between 12-60, with a higher score indicating greater disability (old Oxford score).
Time Frame: 10 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group A MoP | Group B CoC
Number analyzed (Participants) | 29 | 139
score on a scale | 16.4 (5.7) | 18.2 (9.2)

ADVERSE EVENTS:
Time Frame: All adverse events up to 10 years post-op
Description: Definitions according to ISO14155:2013
Arm/Group | Group A MoP | Group B CoC
All-Cause Mortality (participants affected / at risk) | 36/208 | 25/449
Serious Adverse Events (participants affected / at risk) | 63/208 | 89/449
Other Adverse Events (participants affected / at risk) | 1/208 | 2/449
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A MoP (N=208) | Group B CoC (N=449)
Death (General disorders) | 36 (36) | 26 (26) — Death (any cause, not related to procedure/implant)
Device Revision (Surgical and medical procedures) | 15 (15) | 10 (10) — Revision surgery with removal of the study device (any component of the hip)
Dislocation (Musculoskeletal and connective tissue disorders) | 4 (4) | 9 (18) — First and recurrent dislocations
Fracture of femur or acetabulum (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Trochanteric Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Total Knee Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Total Hip replacement contralateral (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Initial cup instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Noise from the hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Heterotopic Ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Facet joint (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain syndrom (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Pain - Intermittent (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Severe hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Deep vein Trombosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aortic Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Sciatic Nerve Encace (Nervous system disorders) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Swelling finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Femoral subsidence (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
BILAT BK AMPUTATIONS (Surgical and medical procedures) | 0 (0) | 1 (1)
Ankle replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Calcar Crack (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Injury after fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Nervous system disorders) | 0 (0) | 1 (1)
Sponteneous bleeds (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Trochanteric Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Thigh Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
vertrebral collapse (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CVA (Vascular disorders) | 0 (0) | 1 (1)
Terminally Ill (General disorders) | 0 (0) | 1 (1)
Pain hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin Discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PSOAS Strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — The initial CRF in the study did not allow to mark an event as serious yes/no. Therefore, all reported events are recorded as an SAE.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A MoP (N=208) | Group B CoC (N=449)
Pain in left lateral thigh after fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fall on shoulder without injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RIGHT CARPAL TUNNEL DECOMPRESSION (Surgical and medical procedures) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Initial CRF in the study did not record if an adverse event was serious yes/no. Where unknown, the event is recorded as serious.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04255394/Prot_SAP_000.pdf